CLINICAL TRIAL: NCT05949047
Title: Biobehavioral Mechanisms of Smartphone-based Cognitive Emotion Regulation Training for Unpaid Primary Caregivers of Persons With Alzheimer's Disease
Brief Title: Smartphone-based Cognitive Emotion Regulation Training for Unpaid Primary Caregivers of Persons With Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bryan Denny (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Bryan Denny, Assistant Professor, William Marsh Rice University
Organization: William Marsh Rice University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY2018-336; 1R01AG074229-01A1 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-07-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Caregivers; Emotions; Emotion Regulation; Stress; Psychological; Psychophysiology
Keywords: emotion regulation; caregiving; affective science; psychophysiology; psychoneuroimmunology
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the "Distancing" group, the "Reinterpretation" group, or a no regulation "Look Only" control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Distancing (Experimental): Participants will receive structured cognitive emotion regulation training from an experimenter during an approximately 10-minute interaction via videoconference in which detailed instructions for implementation of the distancing strategy is explained (i.e. appraising an emotional stimulus as an objective, impartial observer).
  Interventions: Behavioral: Cognitive Emotion Regulation Training via Psychological Distancing
- Reinterpretation (Active Comparator): Participants will receive structured cognitive emotion regulation training from an experimenter during an approximately 10-minute interaction via videoconference in which detailed instructions for implementation of the reinterpretation strategy is explained (i.e. imagining a better outcome than what initially seemed apparent).
  Interventions: Behavioral: Cognitive Emotion Regulation Training via Reinterpretation
- No regulation "Look Only" (No Intervention): The No Regulation "Look Only" Control group will serve as a habituation and natural history control; they will see the same emotional images, but they will only be cued to look and respond naturally for all trials.

INTERVENTIONS:
Behavioral: Cognitive Emotion Regulation Training via Psychological Distancing — The project will randomly assign Alzheimer's Disease or related dementia (AD/ADRD) unpaid primary caregivers to receive a brief course of reappraisal training using either psychological distancing or reinterpretation, or to a no regulation natural history control condition. In the Psychological Distancing group, participants will be asked to down-regulate negative emotion by reappraising an emotional stimulus as an objective, impartial observer.
  Arms: Distancing
Behavioral: Cognitive Emotion Regulation Training via Reinterpretation — The project will randomly assign Alzheimer's Disease or related dementia (AD/ADRD) unpaid primary caregivers to receive a brief course of reappraisal training using either psychological distancing or reinterpretation, or to a no regulation natural history control condition. In the Reinterpretation group, participants will be asked to down-regulate negative emotion by imagining a better outcome (when engaging with an emotional stimulus) than what initially seemed apparent.
  Arms: Reinterpretation

SUMMARY:
Alzheimer's Disease (AD) and Alzheimer's Disease-Related Dementias (ADRD) not only exact a heavy toll on patients, they also impose an enormous emotional, physical, and financial burden on unpaid, often family, caregivers. The strain of providing care for a loved one diagnosed with AD, often across several years, is associated with elevated depression risk and poorer overall health. Emotion regulation skills represent an ideal target for psychological intervention to promote healthy coping in ADRD caregivers. The project seeks to use an experimental medicine approach to test the efficacy and biobehavioral mechanisms of a novel, relatively brief, targeted, scalable, smartphone-based cognitive emotion regulation intervention aimed at improving psychological outcomes (i.e., reducing perceived stress, caregiver burden, and depressive symptoms) in ADRD unpaid primary caregivers as well as examine potential benefits of the caregiver intervention on quality of life in care recipients. Cognitive reappraisal is the ability to modify the trajectory of an emotional response by thinking about and appraising emotional information in an alternative, more adaptive way. Reappraisal can be operationalized via two primary tactics: psychological distancing (i.e. appraising an emotional stimulus as an objective, impartial observer) and reinterpretation (i.e., imagining a better outcome than what initially seemed apparent). The project will investigate the efficacy and underlying biobehavioral mechanisms of a novel, one-week cognitive reappraisal intervention in this population, with follow-up assessments at 2 weeks, 4 weeks, and 3 months. ADRD unpaid primary caregivers will be randomly assigned to receive training in either distancing, reinterpretation, or a no regulation natural history control condition, with ecological momentary assessments of self-reported positive and negative affect, remotely- collected psychophysiological health-related biomarkers (i.e., heart rate variability data) using pre-mailed Polar H10 chest bands, and health-related questionnaire reports. Distancing training is expected to result in longitudinal reductions in self-reported negative affect, longitudinal increases in positive affect, and longitudinal increases in HRV that are larger than those attributable to reinterpretation training and no-regulation control training.

DETAILED DESCRIPTION:
The objective of the research is to use an experimental medicine approach to test the efficacy and biobehavioral mechanisms of a novel, relatively brief, targeted, scalable, smartphone-based cognitive emotion regulation intervention aimed at improving psychological outcomes (i.e., reducing perceived stress, caregiver burden, and depressive symptoms) in unpaid primary caregivers of persons diagnosed with Alzheimer's Disease or a related dementia (ADRD) as well as examine potential benefits of the caregiver intervention on quality of life in care recipients. Cognitive reappraisal (i.e., the ability to modify the trajectory of an emotional response by thinking about and appraising emotional information in an alternative, more adaptive way) represents a highly promising target for psychological intervention in ADRD caregivers. Reappraisal can be operationalized via two primary tactics: psychological distancing (i.e. appraising an emotional stimulus as an objective, impartial observer) and reinterpretation (i.e., imagining a better outcome than what initially seemed apparent). The project builds upon promising preliminary work to investigate the efficacy and underlying biobehavioral mechanisms of a novel, one-week cognitive reappraisal intervention in this population. ADRD unpaid primary caregivers will be randomly assigned to receive training in either distancing, reinterpretation, or a no regulation natural history control condition (Look Only), with one-week of active smartphone-based reappraisal training, with follow-up assessments at 2 weeks, 4 weeks, and 3 months, with longitudinal collection of self-reported positive and negative affect, ecological momentary assessments of daily stress, remotely-collected psychophysiological health-related biomarkers (i.e., heart rate variability data collected using a pre-mailed H10 strap and phone app using bluetooth), and health-related questionnaire reports. The study aims to mechanistically relate changes in psychological and psychophysiological function to prediction of health-relevant behavioral outcomes during a novel emotion regulation intervention never before implemented in this stressed, high risk group.

This research represents a Phase I, Stage I clinical trial. The primary endpoints are the assessments of the psychological and psychophysiological mechanisms mediating behavior change as a function of the cognitive emotion regulation intervention. Psychological mechanisms will be assessed by changes in self-reported positive and negative affect. Psychophysiological mechanisms will be investigated by analysis of heart rate variability data. The secondary endpoint is testing the efficacy of the intervention via assessment of psychological outcomes (i.e., the behavior change, as represented in changes in perceived stress, caregiver burden, and depressive symptoms), as well as care recipient quality of life.

270 ADRD unpaid primary caregivers will be recruited to participate in this study. This research involves random assignment of ADRD caregiver participants to either distancing training, reinterpretation training, or a no regulation natural history control condition (Look Only), as described above, using a parallel intervention model. In particular, the investigators will pseudorandomly assign participants to training groups via initially randomly interspersing 270 condition assignments (90 per cell) and then assigning participants in order accordingly. Male ADRD caregivers as well as caregivers from underrepresented racial and ethnic groups will be oversampled to ensure parity of male and female caregivers as well as equitable representation of underrepresented groups in the sample. Trained experimenters from the study team will administer all 3 conditions (distancing, reinterpretation, and Look Only) with equal frequency. The identity of the experimenter will be incorporated as a covariate during data analysis. Fidelity to the experimental protocol will be maintained via a standardized script for emotion regulation training, modified for each of the three conditions (Distancing, Reinterpretation, Look Only); direct PI training of the Project Coordinator and all research assistants who will acquire data on this protocol; and regular adherence monitoring via ongoing PI observation of Project Coordinator and research assistant training implementation. In addition, the investigators will audiotape training sessions (optionally, via informed consent), with PI review of a randomly-selected 10% of recordings to further ensure fidelity to the protocol.

Power Analyses

Power analysis for caregiver self-reported negative affect:

Sufficient power to assess self-reported negative affect outcomes will be achieved by recruiting 90 participants per training condition. This sample size estimate is based upon a power analysis for detecting an approximate effect size (d = 0.5) previously reported for within and between-subjects behavioral analyses of longitudinal reappraisal training data. Power analyses using this approximate effect size indicate over 95% power (alpha = 0.05) to detect within-group effects and over 90% power (alpha = 0.05) to detect between- group effects should be achieved with 70 participants per condition. Assuming all-cause attrition of 20% (which reflects a liberal upper bound, given past participant attrition rates of approximately 10% in longitudinal studies performed by the current study team), the sample size should provide sufficient power to assess this outcome. Post-attrition, the investigators expect to have analyzable complete data for 72-81 participants per condition.

Power analysis for caregiver heart rate variability (HRV):

Sufficient power to assess respiratory sinus arrhythmia outcomes will be achieved by recruiting 90 participants per training condition. This sample size estimate is based upon a power analysis using an approximate effect size (d = 0.5) previously obtained for within and between-subjects analyses of HRV data. Power analyses using this approximate effect size indicate over 95% power (alpha = 0.05) to detect within- group effects and over 90% power (alpha = 0.05) to detect between-group effects should be achieved with 70 participants per condition. Assuming all-cause attrition of 20% (which reflects a liberal upper bound given past participation attrition rates in longitudinal studies performed by the current study team of approximately 10%), the sample size should provide sufficient power to assess this outcome. Post-attrition, the investigators expect to have analyzable complete data for 72-81 participants per condition.

Power analysis for caregiver perceived stress, caregiver burden, depressive symptoms:

Sufficient power to assess questionnaire outcomes (e.g., perceived stress, caregiver burden, depressive symptoms) will be achieved by recruiting 90 participants per training condition. This sample size estimate is based upon a power analysis using an approximate effect size (d = 0.5) previously reported for within and between-subjects analyses of questionnaire reports measuring these variables (e.g., depressive symptoms; perceived stress). Power analyses using this approximate effect size indicate over 95% power (alpha = 0.05) to detect within-group effects and over 90% power (alpha = 0.05) to detect between-group effects should be achieved with 70 participants per condition. Assuming all-cause attrition of 20% (which reflects a liberal upper bound given past participation attrition rates in longitudinal studies performed by the current study team of approximately 10%), the sample size should provide sufficient power to assess this outcome. Post-attrition, the investigators expect to have analyzable complete data for 72-81 participants per condition.

Power analysis for care recipient affect and quality of life:

Sufficient power to assess care recipient affect and quality of life will be achieved by recruiting 90 participants per training condition. While the precise anticipated effect size for change over time in these care recipient measures as a function of caregiver cognitive emotion regulation training is not known and not expected to be large, a power analysis using a small effect size (d = 0.3) indicates 80% power (alpha = 0.05) to detect within-group effects should be achieved with 71 participants per condition. Assuming all-cause attrition of 20% (which reflects a liberal upper bound given past participation attrition rates in longitudinal studies performed by the current study team of approximately 10%), the sample size should provide sufficient power to assess this outcome. Post-attrition, the investigators expect to have analyzable complete data for 72-81 participants per condition.

Data Analyses

Data analysis will primarily use linear mixed models, incorporating fixed effects for Training Group (Distancing, Reinterpretation, No Regulation Control), Session, and Trial Type (for analyses involving the reappraisal task; Look Neutral, Look Negative, and Reappraise Negative), and their fixed-effect interactions, as well as a random effect consisting of an intercept (main effect) for each participant. In an exploratory follow-up, the investigators will additionally examine models using a random slope per participant. The outcome variables will be changes in self-reported positive and negative affect (via EMA) and HRV (RMSSD) (Aim 1) and changes in health-relevant behavioral outcomes (Aim 2). In these analyses, gender, age, caregiver relationship to care recipient, and baseline caregiving distress burden will be incorporated as covariates. Importantly, the investigators also anticipate having sufficient power to conduct exploratory analyses on the effect of caregiver gender and age on the hypothesized effects (all Aims) given that the investigators will ensure gender balance in each group by oversampling male caregivers (see Recruitment and Retention Plan). This information may help inform future intervention design and assessment (Stage II and beyond) that may arise from the results of this work. Aim 3 will be investigated using multilevel mediation modeling involving training group assignment as the higher-level predictor (X); self-reported positive and negative affect, and HRV data as individual-level mediators (M); and health-relevant behavior as individual-level outcome variables (Y; i.e., a 2-1-1 multilevel mediation model). Relevant covariates indicated above will be incorporated in all mediation models.

Missing data will be imputed using random forest imputation, which mines for complexities (interactions, nonlinearities) in the data while achieving more robust cross-validated prediction of missing-at-random (MAR) data. Loss to follow-up will be mitigated via systematic tracking of participant progress during the experiment (e.g., timeliness and completeness of training via Qualtrics from T1-T7; completion rate for daily EMA pings; and timeliness and completeness of questionnaires). An experimenter will directly contact participants who do not complete study components on schedule (i.e., not completing daily training, responding to fewer than 1 EMA ping per day, or not completing questionnaires on schedule) with reminders about the study schedule and assist with any questions. This checking and reminder system will be in addition to the automated SMS reminders sent via SurveySignal.

ELIGIBILITY:
Inclusion Criteria:

Healthy Adult Caregivers

* Unpaid primary caregiver of patient with Alzheimer's Disease/Alzheimer's Disease and Related Dementias (AD/ADRD)
* At least 18 years of age, with no maximum age, provided that all other inclusion/exclusion criteria are met
* Must be able to speak, read, and write in English
* Must be free of any current or past DSM diagnosis (i.e. healthy adults), with the exception of current or past mood or anxiety disorders or past substance-related disorders (i.e., current or past mood or anxiety disorders and/or past substance-related disorders would not represent an exclusion factor)
* Must have a smartphone. This represents any major iOS or Android-based smartphone. The smartphone will also be used for collection of ecological momentary assessment (EMA) data via SurveySignal.
* Must provide significant level of caregiving to their care recipient
* Must be at least minimally-stressed

Cognitively Impaired Adults

* Must have diagnosed with Alzheimer's Disease/Alzheimer's Disease and Related Dementias (AD/ADRD)
* Must be the care recipient of the primary caregiver who is completing the study
* Must be able to understand and willing to complete a questionnaire and the consent form
* Must have minimum level of dementia symptoms

Exclusion Criteria:

Healthy Adult Caregivers

* Current or past psychiatric disorders (e.g., psychotic and personality disorders) with the exception of current or past mood or anxiety disorders or past substance-related disorders (i.e., current or past mood or anxiety disorders and/or past substance-related disorders would not represent an exclusion factor)
* Currently receiving psychotherapy that specifically addresses caregiver burden/distress or employs cognitive reappraisal as a major component
* Significant visual, auditory, or cognitive impairment that compromises their ability to understand and complete the task
* Caregiver participants who cease meeting inclusion criteria during the study will be dismissed from the study and compensated pro-rata.
* Has formerly participated in a study from our lab involving the same or essentially same design (e.g., former participants who provided pilot/preliminary data for this study)

Cognitively Impaired Adults

* The care recipient does not wish to participate, and/or their caregiver does not want them to participate
* Significant visual, auditory, or cognitive impairment that compromises their ability to understand and complete questionnaires, even with their caregiver's help will exclude them from the study
* Has formerly participated in a study from our lab involving the same or essentially same design (e.g., former participants who provided pilot/preliminary data for this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported negative affect | During Sessions Day 1 - Day 7; this cycle is 7 days
  Self-reported negative affect data collected during completion of emotion regulation task via smartphone
Ecological momentary assessment of positive and negative affect | During Sessions Day 1 - Day 7; this cycle is 7 days
  Ecological momentary assessment (EMA) of positive and negative affect collected during 4 daily afternoon EMA pings via smartphone
Heart rate variability | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Heart rate variability measured via smartphone in conjunction with a Bluetooth-connected H10 Polar Chest Band. Change in heart rate variability assessed at the following timepoints:
Perceived stress | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Perceived stress assessed via the Perceived Stress Scale on a scale of 0 to 4, with 0 indicating "Never" and 4 indicating "Very Often". A higher overall score on the stress scale indicates a worse outcome. Change in self-reports of perceived stress assessed at the following timepoints:
Caregiver burden | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Caregiver burden assessed via the Caregiver Burden Scale on a scale of 0 to 4, with 0 indicating "Never" and 4 indicating "Nearly Always". The greater the total score, the worse the outcome. Change in self-reports of caregiver burden assessed at the following timepoints:
Caregiver quality of life | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Caregiver quality of life assessed via the Caregiver Quality of Life Index on a scale of 0 to 4, with 0 indicating "Not at all" and 4 indicating "Very much". A higher overall score on the Caregiver quality of life index indicates a higher quality of life and better outcome. Change in self-reports of caregiver quality of life assessed at the following timepoints:
Depressive symptoms | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Depressive systems assessed via the Center for Epidemiological Studies-Depression (CES-D) Depression Inventory on a scale of 0 to 3, with 0 indicating "Rarely or none of the time (less than 1 day)," and 3 indicating "Most or all of the time (5-7 days)". The higher the score on the CES-D Depression Inventory, the worse the outcome. Change in self-reports of depressive symptoms assessed at the following timepoints:
Difficulty in regulating emotion | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Difficulty in regulating emotion will be assessed using the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF). There are 5 possible responses to a series of questions: almost never (0-10%), sometimes (11-35%), about half of the time (36-65), most of the time (66%-90%), almost always (91-100%). "Almost never" is the minimum score and "almost always) is the maximum score. Higher scores reflect a worse outcome or greater difficulty with emotion regulation. Change in self-reports of regulating emotions assessed at the following timepoints:
Positive and negative affect | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Positive and negative affect assessed via the Positive and Negative Affect Schedule (PANAS) on a scale of 1 to 5, with a score of 1 indicating "Very slightly or not at all" and a score of 5 indicating "extremely". It is scored using two categories, a positive affect score and a negative affect score. Those with a higher positive affect and lower negative affect score have the most positive outcome. Change in self-reports of positive and negative affect assessed at the following timepoints:
Interpersonal regulation | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Interpersonal regulation efficacy assessed via the Interpersonal Regulation Questionnaire on a scale of 1 to 7, with a score of 1 indicating "strongly disagree" and a scale of 7 indicating "strongly agree". A higher score on this questionnaire indicates a change in self-reports of interpersonal regulation assessed at the following timepoints:
Empathy | Initial training (Day 0), Day 7, Day 14, Day 28, and Month 3
  Empathy Assessed via the Interpersonal Reactivity Index (IRI) on a scale of 0 to 4, with a score of 0 indicating "does not describe me well" and a score of 4 indicating "describes very well". A higher score on this index indicates greater levels of empathy. In this study, the degree of empathy the individual scores does not correlate to a better or worse outcome. The Change in self-reports of empathy assessed at the following timepoints:

SECONDARY OUTCOMES:
Reappraisal usage frequency | Initial training (Day 0)
  General/overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire
Reappraisal usage frequency | Day 7
  General/overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire
Reappraisal usage frequency | Day 14
  General/overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire
Reappraisal usage frequency | Day 28
  General/overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire
Reappraisal usage frequency | Month 3; this period one day long, 3 months after the initial visit)
  General/overall reappraisal usage frequency assessed via the Emotion Regulation Questionnaire
Quick Dementia Rating System (QDRS) | Initial training (Day 0)
  Caregiver-reported assessment of cognitive and behavioral function of care recipients. The QDRS is scored on a continuous scale with a range of 0-30. Higher scores suggest more impairment.
Quick Dementia Rating System (QDRS) | Day 7
  Caregiver-reported assessment of cognitive and behavioral function of care recipients. The QDRS is scored on a continuous scale with a range of 0-30. Higher scores suggest more impairment.
Quick Dementia Rating System (QDRS) | Day 14
  Caregiver-reported assessment of cognitive and behavioral function of care recipients. The QDRS is scored on a continuous scale with a range of 0-30. Higher scores suggest more impairment.
Quick Dementia Rating System (QDRS) | Day 28
  Caregiver-reported assessment of cognitive and behavioral function of care recipients. The QDRS is scored on a continuous scale with a range of 0-30. Higher scores suggest more impairment.
Quick Dementia Rating System (QDRS) | Month 3 (this period is one day long, 3 months after the initial visit)
  Caregiver-reported assessment of cognitive and behavioral function of care recipients. The QDRS is scored on a continuous scale with a range of 0-30. Higher scores suggest more impairment.
Revised Memory and Behavior Problem Checklist (RMBPC) | Month 3 (this period is one day long, 3 months after the initial visit)
  The Revised Memory and Behavior Problem Checklist involves the caregiver a) rating the frequency of observable behavior problems in the dementia patient during the past week (1 = not in the past week, to 4 = daily or more often) and (b) their reaction to each behavior (e.g. how bothered or upset the caregiver feels when the behavior occurs with 0 = not at all to 4 = extremely).
  Frequency Score: The total frequency score is computed to obtain a possible range of 0 to 4, where 0 is the lowest frequency of behavioral problems, and 4 is the highest frequency.
  Reaction Scoring: The total reaction score is computed in the same way, to obtain a possible range of 0 to 4, where 0 as the minimum reaction score (e.g., not being upset about the care recipient's behavioral problems) and 4 as the maximum reaction score (e.g., being extremely upset about the care recipient's behavioral problems).
Care recipient affect | Initial training (Day 0)
  Care recipients will provide valence and arousal ratings by selecting the Self-Assessment Manikin that best exemplifies their emotional state in that moment. Their arousal rating is selected between 9 Manikins that range from a frowning face to a smiling face, with less arousal indicated by a frowning face and greater arousal indicated by a smiling face. Their valence rating is selected between 9 Manikins that range from a small bubble in their chest to a large, protruding bubble in their chest. The lower their valence rating is, the smaller the chest bubble appears. Change in self-reports of valence and arousal assessed at the following timepoints:
Care recipient affect | Day 7
  Care recipients will provide valence and arousal ratings by selecting the Self-Assessment Manikin that best exemplifies their emotional state in that moment. Their arousal rating is selected between 9 Manikins that range from a frowning face to a smiling face, with less arousal indicated by a frowning face and greater arousal indicated by a smiling face. Their valence rating is selected between 9 Manikins that range from a small bubble in their chest to a large, protruding bubble in their chest. The lower their valence rating is, the smaller the chest bubble appears. Change in self-reports of valence and arousal assessed at the following timepoints:
Care recipient affect | Day 14
  Care recipients will provide valence and arousal ratings by selecting the Self-Assessment Manikin that best exemplifies their emotional state in that moment. Their arousal rating is selected between 9 Manikins that range from a frowning face to a smiling face, with less arousal indicated by a frowning face and greater arousal indicated by a smiling face. Their valence rating is selected between 9 Manikins that range from a small bubble in their chest to a large, protruding bubble in their chest. The lower their valence rating is, the smaller the chest bubble appears. Change in self-reports of valence and arousal assessed at the following timepoints:
Care recipient affect | Day 28
  Care recipients will provide valence and arousal ratings by selecting the Self-Assessment Manikin that best exemplifies their emotional state in that moment. Their arousal rating is selected between 9 Manikins that range from a frowning face to a smiling face, with less arousal indicated by a frowning face and greater arousal indicated by a smiling face. Their valence rating is selected between 9 Manikins that range from a small bubble in their chest to a large, protruding bubble in their chest. The lower their valence rating is, the smaller the chest bubble appears. Change in self-reports of valence and arousal assessed at the following timepoints:
Care recipient affect | Month 3 (this period is one day long, 3 months after the initial visit)
  Care recipients will provide valence and arousal ratings by selecting the Self-Assessment Manikin that best exemplifies their emotional state in that moment. Their arousal rating is selected between 9 Manikins that range from a frowning face to a smiling face, with less arousal indicated by a frowning face and greater arousal indicated by a smiling face. Their valence rating is selected between 9 Manikins that range from a small bubble in their chest to a large, protruding bubble in their chest. The lower their valence rating is, the smaller the chest bubble appears. Change in self-reports of valence and arousal assessed at the following timepoints:
Care recipient quality of life | Initial training (Day 0)
  Care recipients will rate their quality of life using the Quality of Life in Alzheimer's Disease Scale (QoL-AD). There are 4 possible responses to a series of questions: poor, fair, good, and excellent. "Poor" is the minimum score and "excellent" is the maximum score. Higher scores mean a better outcome or greater quality of life. Change in self-reports of care recipient quality of life at the following timepoints:
Care recipient quality of life | Day 7
  Care recipients will rate their quality of life using the Quality of Life in Alzheimer's Disease Scale (QoL-AD). There are 4 possible responses to a series of questions: poor, fair, good, and excellent. "Poor" is the minimum score and "excellent" is the maximum score. Higher scores mean a better outcome or greater quality of life. Change in self-reports of care recipient quality of life at the following timepoints:
Care recipient quality of life | Day 14
  Care recipients will rate their quality of life using the Quality of Life in Alzheimer's Disease Scale (QoL-AD). There are 4 possible responses to a series of questions: poor, fair, good, and excellent. "Poor" is the minimum score and "excellent" is the maximum score. Higher scores mean a better outcome or greater quality of life. Change in self-reports of care recipient quality of life at the following timepoints:
Care recipient quality of life | Day 28
  Care recipients will rate their quality of life using the Quality of Life in Alzheimer's Disease Scale (QoL-AD). There are 4 possible responses to a series of questions: poor, fair, good, and excellent. "Poor" is the minimum score and "excellent" is the maximum score. Higher scores mean a better outcome or greater quality of life. Change in self-reports of care recipient quality of life at the following timepoints:
Care recipient quality of life | Month 3 (this period is one day long, 3 months after the initial visit)
  Care recipients will rate their quality of life using the Quality of Life in Alzheimer's Disease Scale (QoL-AD). There are 4 possible responses to a series of questions: poor, fair, good, and excellent. "Poor" is the minimum score and "excellent" is the maximum score. Higher scores mean a better outcome or greater quality of life. Change in self-reports of care recipient quality of life at the following timepoints:

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Denny, Ph.D., Principal Investigator — William Marsh Rice University
Locations (1):
- Rice University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Pursuant to the NIH Data Sharing Policy, we have created a Data Sharing Plan for the project. Under this plan, and pursuant to IRB regulations at Rice University and Baylor College of Medicine, fully de-identified raw data (defined below) will be made publicly available through the mechanisms below after the analysis process is complete and research manuscript(s) are finalized. Available data will include a compendium of de-identified training condition assignments; raw (i.e. individual subject-by-condition level) negative affect self-reports; ecological momentary assessment (EMA) reports; questionnaire data; and raw heart rate variability data. All datafiles will be uploaded to the Open Science Framework, a free, open-science data repository.
Supporting Information: Study Protocol
Time Frame: De-identified data will be made available after the analysis process is complete and research manuscripts are finalized. There is no fixed end date for data access.
Access Criteria: Data will be publicly available on the Open Science Framework (https://osf.io), a free, open-science data repository.

REFERENCES:
- [Background] Denny BT, Ochsner KN. Behavioral effects of longitudinal training in cognitive reappraisal. Emotion. 2014 Apr;14(2):425-33. doi: 10.1037/a0035276. Epub 2013 Dec 23. PMID 24364856
- [Background] Denny BT. Getting better over time: A framework for examining the impact of emotion regulation training. Emotion. 2020 Feb;20(1):110-114. doi: 10.1037/emo0000641. PMID 31961188
- [Background] Butler, M., J.E. Gaugler, K.M.C. Talley, H.I. Abdi, P.J. Desai, S. Duval, M.L. Fort, V.A. Nelson, W. Ng, J.M. Ouellette, E. Ratner, J. Saha, T. Shippee, B.L. Wagner, T.J. Wilt, and L. Yeshi, Care Interventions for People Living With Dementia and Their Caregivers. Comparative Effectiveness Review No. 231. (Prepared by the Minnesota Evidence-based Practice Center under Contract No. 290-2015- 00008-I.) AHRQ Publication No. 20-EHC023. 2020: Rockville, MD.
- [Background] Brewster P, Barnes L, Haan M, Johnson JK, Manly JJ, Napoles AM, Whitmer RA, Carvajal-Carmona L, Early D, Farias S, Mayeda ER, Melrose R, Meyer OL, Zeki Al Hazzouri A, Hinton L, Mungas D. Progress and future challenges in aging and diversity research in the United States. Alzheimers Dement. 2019 Jul;15(7):995-1003. doi: 10.1016/j.jalz.2018.07.221. Epub 2018 Sep 19. PMID 30240574
- [Background] Boots LM, de Vugt ME, van Knippenberg RJ, Kempen GI, Verhey FR. A systematic review of Internet-based supportive interventions for caregivers of patients with dementia. Int J Geriatr Psychiatry. 2014 Apr;29(4):331-44. doi: 10.1002/gps.4016. Epub 2013 Aug 20. PMID 23963684
- [Background] Schulz R. The Future of Caregiver Efficacy Research: Commentary on "Long-Term Outcomes of the Benefit-Finding Group Intervention for Alzheimer Family Caregivers". Am J Geriatr Psychiatry. 2019 Sep;27(9):995-997. doi: 10.1016/j.jagp.2019.04.001. Epub 2019 Apr 10. No abstract available. PMID 31031074
- [Background] Godwin KM, Mills WL, Anderson JA, Kunik ME. Technology-driven interventions for caregivers of persons with dementia: a systematic review. Am J Alzheimers Dis Other Demen. 2013 May;28(3):216-22. doi: 10.1177/1533317513481091. Epub 2013 Mar 25. PMID 23528881
- [Background] Berking M, Ebert D, Cuijpers P, Hofmann SG. Emotion regulation skills training enhances the efficacy of inpatient cognitive behavioral therapy for major depressive disorder: a randomized controlled trial. Psychother Psychosom. 2013;82(4):234-45. doi: 10.1159/000348448. Epub 2013 May 22. PMID 23712210
- [Background] Berking M, Wupperman P, Reichardt A, Pejic T, Dippel A, Znoj H. Emotion-regulation skills as a treatment target in psychotherapy. Behav Res Ther. 2008 Nov;46(11):1230-7. doi: 10.1016/j.brat.2008.08.005. Epub 2008 Aug 30. PMID 18835479